CLINICAL TRIAL: NCT04306783
Title: In-Home Sensor Monitoring of Older Adults With Cancer: A Pilot Study
Brief Title: In-Home Sensor Monitoring of Older Adults With Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator is leaving the university
Sponsor: Washington University School of Medicine (Other)
Collaborators: Institute of Clinical and Translational Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202001189
Record Dates: First submitted 2019-11-05; First posted 2020-03-13 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: In-Home Sensor Monitoring (Experimental): Older adults with cancer undergoing systemic cancer treatment will undergo passive monitoring with motion sensors and bed sensor. Passive infrared (PIR) motion sensors will be installed in their homes to detect presence in a particular room (e.g., bathroom or kitchen) as well as for specific activities. There will also be a bed sensor, which is a pneumatic strip installed under the bed linens, which measures displacement of the resident's upper torso as he or she lies on the bed. Participants will complete a baseline primarily self-administered survey, an abbreviated assessment with each follow up clinic visit (at least once per month) for 6 months of follow up and a final end of study assessment.
  Interventions: Other: In-home sensor monitoring
- Arm B: Survey Only (No Intervention): Patients that choose to not proceed with in-home sensor monitoring will be asked to complete a brief survey that explores attitudes regarding in-home sensor monitoring

INTERVENTIONS:
Other: In-home sensor monitoring — -Installed and maintained by Foresite Healthcare
  Arms: Arm A: In-Home Sensor Monitoring

SUMMARY:
The investigators propose a pilot study of monitoring a sample of 6 older patients receiving active cancer treatment over a period of 6 months with in-home sensor monitors installed and maintained by Foresite Healthcare. The investigators also propose exploring the beliefs and attitudes of those who are not willing to allow in-home sensor monitoring by asking them to complete a brief survey related to in-home sensor monitoring. The investigators hypothesize that patients will find the equipment acceptable and unintrusive, that changes in home-monitored patient parameters will precede clinical events and that patient trajectories will be more fully characterized with the in home sensors.

ELIGIBILITY:
Inclusion Criteria:

Arm A:

* Age ≥ 65
* Receiving systemic cancer therapy, including conventional chemotherapy, novel/targeted agents OR will begin systemic therapy within the next 4 weeks.
* Estimated life expectancy >1 year
* Anticipated to receive ongoing care at Siteman Cancer Center and its satellite sites
* Willing to have sensors installed in 1-2 primary living areas (e.g. living room and bedroom)
* Continuous home internet connection
* Able to understand and willing to sign an IRB-approved written informed consent document

Arm B:

* Age ≥ 65
* Receiving systemic cancer therapy, including conventional chemotherapy, novel/targeted agents OR will begin systemic therapy within the next 4 weeks.
* Estimated life expectancy >1 year
* Anticipated to receive ongoing care at Siteman Cancer Center and its satellite sites
* Able to understand and willing to sign an IRB-approved written informed consent document

Exclusion Criteria:

Arm A:

* Inability to read and understand English
* Only receiving hormonal agents (e.g. anti-estrogen or anti-androgen)
* Lives in institutional setting where instrumental activities of daily living are completed for patient by paid staff

Arm B:

* Inability to read and understand English
* Only receiving hormonal agents (e.g. anti-estrogen or anti-androgen)
* Lives in institutional setting where instrumental activities of daily living are completed for patient by paid staff

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of in-home sensor monitoring as measured by a modified version of the Intelligent Systems for Assessment of Aging Technology Survey (Arm A only) | 6 months
  * 11 questions about how the participant would feel about in-home sensor monitoring, the participant can choose from 1 = strongly agree to 5 = strongly disagree. A higher score means the participant that does not feel comfortable with in-home sensor monitoring
  * 2 questions about concerns about information gathered by the in-home sensor monitoring might be shared, answers range from 1 = very concerned to 4 = not concerned at all. A higher score indicates participants are uncomfortable with sharing of in-home sensor monitoring data.
  * 4 questions about the participants experience with in-home sensor monitoring, the participant can choose from 1 = strongly agree to 5 = strongly disagree. A lower score indicates that the participant feels like in-home sensor monitoring interferes with their daily activities.
Heart rate (Arm A only) | 6 months
  -A meaningful change is heart rate outside the normal range of 60-100
Changes in gait speed of .1m/s or more (Arm A only) | 6 months
Stride length (Arm A only) | 6 months
Number of Falls (Arm A only) | 6 months
Number of Hospitalizations (Arm A only) | 6 months
Number of Emergency room visits (Arm A only) | 6 months
Number of Infections requiring medical intervention (e.g. oral antibiotics) (Arm A only) | 6 months
Number of grade ≥3 adverse events measured by CTCAE (Arm A only) | 6 months
Patient reported outcomes of 10 common symptoms (Arm A) | 6 months
  * The reported symptoms are decreased appetite, pain, decreased activity level, depressed mood, nausea, vomiting, diarrhea, constipation, shortness of breath, and insomnia
  * Patient reports on a scale of 1-5 with 1 indicating the symptom is absent and 5 indicating the symptom is severe
Reason for not choosing in-home monitoring as measured by a modified version of the Intelligent Systems for Assessment of Aging Changes Technology Survey (Arm B only) | At the time of invitation to participate in the study (Day 1)
  * 11 questions about how the participant would feel about in-home sensor monitoring, the participant can choose from 1 = strongly agree to 5 = strongly disagree. A higher score means that the participant that does not feel comfortable with in-home sensor monitoring
  * 2 questions about concerns about information gathered by the in-home sensor monitoring might be shared, answers range from 1 = very concerned to 4 = not concerned at all. A higher score indicates participants are uncomfortable with sharing of in-home sensor monitoring data.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya M Wildes, M.D., MSCI, Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu